CLINICAL TRIAL: NCT00974233
Title: Phase II Study of Bendamustine and Rituximab Induction Chemoimmunotherapy With Maintenance Lenalidomide and Rituximab in Relapsed/Refractory CLL/SLL
Brief Title: Study of Bendamustine/Rituxan Induction Chemotherapy With Revlimid Maintenance for Relapsed/Refractory CLL and SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO08405; RV-CLL/SLL-PI-397; A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); H-2009-0087 (Other: Institutional Review Board); NCI-2011-00646 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2017-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction/Maintenance chemotherapy (Experimental): Bendamustine + rituximab induction therapy followed by lenalidomide maintenance therapy
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bendamustine — 90 mg/m2/day IV days 1 and 2 every 28 days for 6 cycles
  Other Names: Treanda
Drug: Rituximab — 375 mg/m2 Day 1 every 28 days for 6 cycles
  Other Names: rituxan
Drug: Lenalidomide — 5 mg/day days 1-28 of each 28 day cycle, up to 12 cycles maximum. Dose escalation to 10 mg/day allowed after one cycle as defined in the protocol.
  Other Names: revlimid; CC-5013

SUMMARY:
The purpose of this research is to evaluate a new combination of chemotherapy drugs for CLL/SLL using the drugs bendamustine (an intravenous chemotherapy drug), rituximab (an intravenous medication called a monoclonal antibody), and lenalidomide (an anti-cancer pill).

The purpose of this study is to see if giving the chemotherapy pill lenalidomide after treatment with bendamustine and rituximab is able to prolong the period of time before the cancer starts growing again and causing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed,CLL/SLL, documented relapsed or refractory disease after at least one prior chemotherapy regimen.
* In cases of SLL, patients must have at least one bidimensionally measurable lesion at least ≥1.5 cm measured in one dimension.
* ECOG performance status of 0-2 at study entry
* Laboratory test results within these ranges: ANC <=1500/μL, Platelet count <= 100,000/μL. Patients with ANC <1500/μL or plt <100,000/μL with splenomegaly or extensive bone marrow involvement as the etiology for their cytopenias are eligible.
* creatinine clearance of >60 mL/min as determined by the Cockcroft-Gault calculation.
* Total bilirubin <= 2X upper limit laboratory normal (ULN). Patients with non-clinically significant elevations of bilirubin due to Gilbert's disease are not required to meet these criteria.
* Serum transaminases AST (SGOT) and ALT (SGPT) <=5x ULN, Serum alkaline phosphatase ≤5 X ULN.
* Disease free of prior malignancies for ≥ 2 years with the exception of basal or squamous cell skin carcinoma, carcinoma "in situ" of the breast or cervix, or localized prostate cancer (treated definitively with hormone therapy, radiotherapy, or surgery).
* Patients may have received prior therapy with bendamustine or lenalidomide, but must not have disease that is refractory to bendamustine or lenalidomide.
* Prior therapy with rituximab is permitted, even in the setting of rituximab refractory disease.

Exclusion Criteria:

* Has received >5 lines of prior therapy for their disease. Re-treatment with an identical regimen does not count as a new regimen.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form or comply with the protocol treatment.
* Pregnant or breast feeding females. Lactating females must agree not to breast feed while taking lenalidomide.
* Prior history or current evidence of central nervous system or leptomeningeal involvement.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known to be positive for HIV or infectious hepatitis, type B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Chang, MD, Principal Investigator — University of Wisconsin, Madison
Locations (10):
- United States (10):
  - St Vincent Regional Cancer Center, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Mercy Health System Heme/Onc, Janesville, Wisconsin
  - Gundersen Clinic, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Chang JE, Wang T, Kim K, Folstad M, Endres M, Howard M, Kenkre V, Fletcher C, Rajguru S. Maintenance low-dose fixed duration lenalidomide and rituximab following bendamustine and rituximab induction in previously untreated chronic lymphocytic leukemia and small lymphocytic lymphoma. Leuk Lymphoma. 2024 Oct;65(10):1456-1464. doi: 10.1080/10428194.2024.2360535. Epub 2024 Jun 10. PMID 38856101
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Research subjected from the University of Wisconsin and 7 Wisconsin Oncology Network institutions were enrolled from October 2009 to November 2011. Subjects were enrolled from outpatient hematology clinics at each participating institution.
Groups:
- Induction Chemoimmunotherapy + Maintenance Lenalidomide: Induction therapy: Bendamustine 90 mg/m2 IV on days 1 & 2 + rituximab 375 mg/m2 IV on day 1 (permitted on day 2 of cycle 1) every 28 days for total of 6 treatment cycles. Maintenance therapy: Lenalidomide 5-10 mg orally continuously of each 28-day cycles for total of 12 treatment cycles.
Period: Induction Chemoimmunotherapy
Arm/Group | Induction Chemoimmunotherapy + Maintenance Lenalidomide
Started | 34
Completed | 19
Not Completed | 15
Not completed — Death | 2
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Period: Maintenance Lenalidomide
Arm/Group | Induction Chemoimmunotherapy + Maintenance Lenalidomide
Started | 19
Completed | 6
Not Completed | 13
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 8

BASELINE CHARACTERISTICS:
Population: Subjects with progressive chronic lymphocytic leukemia/small lymphocytic lymphoma receiving 1-5 prior unique treatment regimens.
Groups:
- Overall Study Population: Patient population with chronic lymphocytic leukemia/small lymphocytic lymphoma with progressive disease in need of therapy after at least 1 prior chemotherapy regimen, but no more than 5 prior unique chemotherapy regimens (retreatment with identical regimen did not count as a unique regimen).
Arm/Group | Overall Study Population
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 67 [48 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
ECOG performance status [Number; unit: participants] — ECOG performance status (PS) evaluated clinically in all patients on a scale from 0-5, with higher ECOG PS indicating worse functional impairment (i.e., ECOG PS of zero = asymptomatic, fully functional patient; ECOG PS of 5 = death).
  participants
    ECOG performance status 0-1 | 32
    ECOG performance status 2 | 2
Disease staging [Number; unit: participants] — Rai staging is a clinical evaluation taking into account blood counts and physical exam findings, with staging ranging from 0-4 (more advanced staging corresponding with higher numbers).
  Ann Arbor staging is an evaluation of physical exam finding combined with imaging evaluation (usually CT imaging) to determine extent of lymph node enlargement, with staging ranging from 1-4 (more advanced staging corresponding with higher numbers).
  participants
    Rai stage 1/2 (CLL) | 12
    Rai stage 3/4 (CLL) | 14
    Ann Arbor stage 1/2 (SLL) | 1
    Ann Arbor 3/4 (SLL) | 7
Median prior therapies [Median (Full Range); unit: prior therapies] — Describes number of unique prior therapies received by subjects, including monoclonal antibody therapy (i.e., single-agent rituximab) or cytotoxic chemotherapy-based therapies. Retreatment with an identical regimen was not counted as a unique therapy. Subjects required at least one cytotoxic chemotherapy-based therapy for eligibility.
  prior therapies | 2 [1 to 4]
Prior therapy with fludarabine [Number; unit: participants]
  Prior fludarabine-based therapy | 23
  No previous fludrarabine exposure | 11
Refractory to most recent therapy [Number; unit: participants]
  Refractory to most recent therapy | 4
  Not refractory to most recent therapy | 30
Elevated serum lactate dehydrogenase (LDH) level [Number; unit: participants] — Lactate dehydrogenase (LDH) is associated with cell growth and turnover in the body. Higher levels of LDH tend to be associated with more rapid tumor growth and is a marker of higher risk lymphoma/leukemia.
  participants
    Enrollment LDH elevated | 20
    Enrollment LDH not elevated | 14
Baseline cytogenetics [Number; unit: participants]
  17p or 11q deletions | 11
  13q deletion | 2
  Trisomy 12 | 8
  Normal | 3
  Unknown | 10
Prior therapy with rituximab [Number; unit: participants]
  Prior therapy with rituximab | 27
  No prior therapy with rituximab | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary endpoint of this study was progression-free survival (PFS), defined as the number of days from the day of first study drug administration to the day the patient experienced disease progression or death from any cause. Response and progression in cases of small lymphocytic lymphoma(SLL) were evaluated using the International Working Group Criteria for response in NHL (Cheson, et al 1996). Response and progression in cases of chronic lymphocytic leukemia (CLL) were evaluated using the NCI-sponsored CLL Working Group guidelines for CLL (Cheson, et al 2007).
Time Frame: 42 months (6 months induction therapy, 12 months maintenance, 24 months long-term follow-up)
Population: The study was designed to test the null hypothesis that the median PFS with induction BR and maintenance lenalidomide is at most 18 months versus the alternative hypothesis that median PFS is >18 months, at a one-sided significance level of 0.10 with a power of 80%.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction/Maintenance Chemotherapy
Number analyzed (Participants) | 34
months | 18.3 [10.6 to 24.3]

2. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from the day of first study drug administration until progression of CLL/SLL or death from any cause. PFS is reported as the proportion of participants with PFS up to 42 months.
Time Frame: 42 months (6 months induction therapy, 12 months maintenance, 24 months long-term follow-up)
Measure: Median (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Induction/Maintenance Chemotherapy
Number analyzed (Participants) | 34
Proportion of participants
  1-year progression-free survival | 0.62 [0.47 to 0.80]
  2-year progression-free survival | 0.35 [0.22 to 0.56]
  3-year progression-free survival | 0.23 [0.12 to 0.43]

3. Secondary Outcome: Objective Response Rate (Complete + Partial Responses)
Description: Response and progression in cases of SLL were evaluated using the International Working Group Criteria for response in NHL (Cheson, et al 1996). Response and progression in cases of CLL were evaluated using the NCI-sponsored CLL Working Group guidelines for CLL (Cheson, et al 2007). Complete response defined as resolution enlarged lymph nodes, spleen and liver; normalization of blood counts (neutrophils, hemoglobin, platelets); no residual CLL/SLL detectable in the bone marrow. Partial response defined as 50% or more reduction in size of enlarged lymph nodes, liver or spleen; 50% or more improvement of blood counts; 50% or more improvement in the blood lymphocyte count. Progressive disease defined as 50% or more increase in the combined measurements of at least 2 lymph nodes as measured on CT scans or the appearance of new enlarged lymph nodes; 50% of more increase in the size of the spleen or liver; 50% or more increase in blood lymphocyte count.
Time Frame: 42 months (6 months induction therapy, 12 months maintenance, 24 months long-term follow-up)
Measure: Number; unit: participants
Groups:
- Complete Response (CR): Complete response defined as resolution enlarged lymph nodes, spleen and liver; normalization of blood counts (neutrophils, hemoglobin, platelets); no residual CLL/SLL detectable in the bone marrow.
- Partial Response (PR): Partial response defined as 50% or more reduction in size of enlarged lymph nodes, liver or spleen; 50% or more improvement of blood counts; 50% or more improvement in the blood lymphocyte count.
- Stable Disease: Stable disease includes cases where there has been objective improvement in blood counts and lymph node size, but does not meet criteria for either a complete or partial response.
- Overall Response Rate: Includes complete and partial responses.
Arm/Group | Complete Response (CR) | Partial Response (PR) | Stable Disease | Overall Response Rate
Number analyzed (Participants) | 34 | 34 | 34 | 34
participants | 7 | 12 | 9 | 19

4. Secondary Outcome: Toxicities Observed With Induction Chemotherapy and Maintenance Therapy
Description: Toxicities were reported using the Common Terminology Criteria for Adverse Events, version 3.0.
Time Frame: 42 months (6 months induction therapy, 12 months maintenance, 24 months long-term follow-up)
Population: Toxicities were reported using the Common Terminology Criteria for Adverse Events, version 3.0.
Measure: Number; unit: participants
Groups:
- Induction Chemoimmunotherapy: Bendamustine 90 mg/m2 IV on days 1 & 2 + rituximab 375 mg/m2 IV on day 1 (permitted on day 2 of cycle 1) every 28 days for total of 6 treatment cycles.
- Maintenance: Lenalidomide 5-10 mg administered orally daily as continuous therapy for up to 12 treatment cycles (28-day treatment cycles) in patients without disease progression or treatment-related toxicities that would prohibit ongoing treatment.
Arm/Group | Induction Chemoimmunotherapy | Maintenance
Number analyzed (Participants) | 34 | 19
participants
  Grade 3 leukopenia | 5 | 6
  Grade 4 leukopenia | 5 | 1
  Grade 3 neutropenia | 6 | 7
  Grade 4 neutropenia | 14 | 2
  Grade 3 anemia | 1 | 0
  Grade 3 thrombocytopenia | 5 | 1
  Grade 4 thrombocytopenia | 2 | 0
  Grade 3 febrile neutropenia | 4 | 1
  Grade 3 infection | 10 | 4
  Grade 4 infection | 1 | 1
  Grade 5 infection | 1 | 0
  Grade 3 fatigue | 2 | 0
  Grade 4 fatigue | 0 | 1
  Grade 3 nausea/emesis | 3 | 0
  Grade 3 serum transaminase levels (Gr 3/Gr 4) | 4 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the day of first study drug administration until death from any cause.
Time Frame: 42 months (6 months induction therapy, 12 months maintenance, 24 months long-term follow-up)
Population: Overall survival (OS) was measured for all enrolled subjects as the time from the day of first study drug administration until death from any cause.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Study Population
Number analyzed (Participants) | 34
months | 42.8 [33.7 to 69.5]

ADVERSE EVENTS:
Time Frame: Adverse event date was captured from the time of study enrollment until at least 30 days following the final dose of study treatment.
Description: Any serious or unexpected adverse event was reported during the entire duration of long-term follow-up.
Arm/Group | Induction Chemoimmunotherapy | Maintenance
Serious Adverse Events (participants affected / at risk) | 14/34 | 8/19
Other Adverse Events (participants affected / at risk) | 34/34 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Chemoimmunotherapy (N=34) | Maintenance (N=19)
Grade 4 neutropenia (Blood and lymphatic system disorders) | 14 (14) | 2 (2) — SAEs included any grade 2-3 unexpected event with at least probable attribution, grade 4-5 toxicity regardless of attribution. Number of events includes worst grade toxicity per patient.
Grade 3 neutropenia (Blood and lymphatic system disorders) | 6 (6) | 7 (7) — Includes all events of grade 3 neutropenia, regardless of whether or not resulted in hospitalization of other definition of SAE.
Grade 4 thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Includes all events of grade 4 thrombocytopenia, as required by definition of SAE per protocol.
Grade 3 thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) — Includes all events of grade 3 thrombocytopenia, regardless of whether or not resulted in hospitalization of other definition of SAE.
Grade 4 leukopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) — Includes all events of grade 4 leukopenia, as defined by SAE reporting per protocol.
Grade 3 leukopenia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) — Includes all events of grade 3 leukopenia, regardless of whether or not resulted in hospitalization of other definition of SAE.
Grade 4 febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0)
Grade 3 febrile neutropenia (Infections and infestations) | 4 (4) | 1 (1)
Grade 5 infections (Infections and infestations) | 1 (1) | 0 (0)
Grade 4 infections (Infections and infestations) | 1 (1) | 1 (1)
Grade 3 tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Grade 3 thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — Includes events that occurred during treatment and during long-term follow-up phase of treatment.
Grade 3 prolonged QTc interval (Cardiac disorders) | 0 (0) | 1 (1)
Grade 5 heart failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Chemoimmunotherapy (N=34) | Maintenance (N=19)
Grade 3 Infections (Infections and infestations) | 10 (10) | 4 (4) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 3 fatigue (General disorders) | 2 (2) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 fatigue (General disorders) | 0 (0) | 6 (6) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 3 emesis (Gastrointestinal disorders) | 2 (2) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 3 diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 3 hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 3 elevated AST/ALT (Hepatobiliary disorders) | 4 (4) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 AST/ALT (Hepatobiliary disorders) | 4 (4) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 night sweats (General disorders) | 0 (0) | 3 (3) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 headache (Nervous system disorders) | 0 (0) | 3 (3)
Grade 1-2 musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 3 pain NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 1-2 emesis (Gastrointestinal disorders) | 2 (2) | 1 (1) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.
Grade 2 stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) — Worst grade toxicity per patient. Includes toxicities that are expected and not meeting other criteria for serious per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No